CLINICAL TRIAL: NCT05691231
Title: Long-Term Assessment of the Safety and Performance of the NuVasive Simplify Disc at Two Levels
Status: Enrolling by invitation | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.TDR1022
Record Dates: First submitted 2023-01-11; First posted 2023-01-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cervical Disc Disease; Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Simplify Disc: Extended follow-up of subjects treated with the Simplify Disc during IDE study NCT03123549 and followed in the post-approval study NCT04980378.
  Interventions: Device: NuVasive Simplify Cervical Artificial Disc

INTERVENTIONS:
Device: NuVasive Simplify Cervical Artificial Disc — Simplify Disc is a weight-bearing cervical artificial disc implant consisting of PEEK (polyetheretherketone) endplates and one semi-constrained, fully articulating, mobile Zirconia Toughened Alumina ceramic (ZTA) core.

SUMMARY:
A prospective, multicenter post-market clinical follow-up study to evaluate the 10-year long-term safety and effectiveness of the Simplify Disc at two levels in subjects who were enrolled in the IDE study (NCT03123549) and/or post approval study (NCT04980378).

ELIGIBILITY:
Inclusion Criteria:

1. Subject was enrolled in the Simplify Disc IDE (NCT03123549) and/or PAS (NCT04980378) at a participating study site
2. Patient understands the conditions of enrollment and is willing sign an informed consent form to participate in the study

Exclusion Criteria:

1. Subject had an SSI at the index level during the IDE study (NCT03123549) or the PAS (NCT04980378)
2. Subject was withdrawn or withdrew consent to participate in the IDE study (NCT03123549) or PAS (NCT04980378)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes subjects treated with the NuVasive Two Level Simplify Disc in IDE study (NCT03123549) and followed in the PAS (NCT04980378).
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2029-02-10 (Estimated); Study Completion 2029-05-10 (Estimated)

PRIMARY OUTCOMES:
Clinical Composite Success Rate | 10 years
  Individual success is defined as at least a 15 point improvement in Neck Disability Index (NDI) Score at 120 months compared with baseline, maintenance or improvement in neurologic status at 120 months compared with baseline, no additional surgical procedure at the index level within 120 months, and the absence of a serious adverse event classified as implant-associated or implant/surgical procedure-associated within 120 months. A subject must meet each criterion to be considered an overall study success.
  NDI scale is reported in a range from 0 - 100, with 0 consistent with best ability to function and 100 with worst ability to function.

SECONDARY OUTCOMES:
Percentage of subjects meeting the minimal clinically important difference (MCID) for NDI at each annual timepoint | 10 years
  Neck Disability Index; scale is reported in a range from 0-100, with 0 consistent with best ability to function and 100 worst ability to function.
Percentage of subjects meeting MCID for neck and arm pain questionnaire for each of the following pain locations: neck pain, arm pain, left arm pain, right arm pain. | 10 years
  Neck and arm pain questionnaire, scale is reported in a range from 0 to 10, with 0 consistent with no pain and 10 with most pain
Motor status at each annual timepoint compared to baseline | 10 years
  A change of one or more grade levels in muscle strength will be regarded as clinically significant.
Sensory status at each annual timepoint compared to baseline | 10 years
  Sensation will be graded as normal or abnormal (diminished or absent). Any changes from abnormal to normal or absent to diminished will be regarded as clinically significant improvement.
SF-36® Health Survey at each annual timepoint compared to baseline | 10 years
  The SF-36 is a multipurpose survey with 36 questions. The questions were combined, scored and weighted to create mental and physical functioning and overall health-related quality of life. Higher scores indicate better outcomes. Scores range from 0-100.
Dysphagia Handicap Index1 (DHI) at each annual timepoint compared to baseline | 10 years
  DHI is scored from 0-100, with a higher score indicative of a less desirable outcome.
Disc height at each annual timepoint will be compared to baseline | 10 years
  Average disc height is calculated as the simple average of the anterior and posterior disc heights
Adjacent level disc degeneration (ALDD) at each annual timepoint will be compared to baseline | 10 years
  ALDD is graded in accordance with definitions adapted from Kellgren and Lawrence: None; Doutbtful;Minimal;Moderate;Severe
Displacement or migration of the Simplify Disc at each annual timepoint will be compared to the post-op timepoint in the IDE study (NCT03123549) | 10 years
  Device migration assesses significant movement of the implant postoperatively. Changes of >3 mm will be considered significant due to the margin of error in radiographic determination of displacement distances.
Range of motion (ROM) at each annual timepoint compared to baseline | 10 years
  Changes in Global Range of Motion will be calculated by subtracting the range of motion measured at one time point from the baseline range of motion. Change in Global Range of Motion will be reported in units of degrees.
Rate of adverse events attributable to Simplify Disc, or use of additional NuVasive instruments, implants, or technologies at each annual timepoint | 10 years
  Number of adverse events related to Simplify Disc or additional NuVasive products
Patient satisfaction and perceived effect at each annual timepoint | 10 years
  Patient questionnaire assessing satisfaction with treatment and perceived effect of treatment. Success for each satisfaction question will be defined as either a "Definitely True" or "Mostly True" response. Success for the perceived effect question will be defined as either a "Completely Recovered," "Much Improved," or "Slightly Improved" response.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, Study Director — NuVasive
Locations (2):
- United States (2):
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - Texas Back Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No